CLINICAL TRIAL: NCT02467751
Title: Metabolic Profile in Women of Different Body Composition With Polycystic Ovary Syndrome
Brief Title: Women With Polycystic Ovary Syndrome (PCOS)
Acronym: PCOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Principal Investigator, Carolina Furtado Macruz, Doctor, Irmandade da Santa Casa de Misericordia de Sao Paulo
Other Study IDs: 167/10
Record Dates: First submitted 2015-03-25; First posted 2015-06-10 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Metabolic profile in women of different body composition with polycystic ovary syndrome.

DETAILED DESCRIPTION:
Will be performed case-control study with women with Polycystic Ovary Syndrome, according to the Rotterdam criteria and body mass index between 18 to 29.9. The control group will consist of women without Polycystic Ovary Syndrome, with a body mass index of 18 to 29.9 and no other comorbidities. In both groups collect anthropometric data such as age, weight, height, waist circumference and blood pressure. Exams will be requested: metabolic profile (total cholesterol (mg/dL) and fractions, triglycerides (mg/dL), blood count, liver function (U/L) and classical glycemic index (mg/dL); hormonal profile - insulin (uIU/ml), luteinizing hormone (IU/L), follicle stimulating hormone (IU/L), thyreostimulating hormone (uIU/ML), total and free testosterone (ng/ml), 17-hydroxyprogesterone (ng/ml), dehydroepiandrosterone (ng/ml), prolactin (ug/ml). Body composition (BMI) will be performed by absorption technique of two low energy beams emitted by X-ray - full body densitometry (DEXA). Expected result: To evaluate visceral fat and truncal of patients with diagnosis of Polycystic Ovary Syndrome without obesity.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic Ovary Syndrome , body mass index of 18 to 29.9, without contraceptive use.

Exclusion Criteria:

* Hypothyroidism, hyperprolactinaemia (defined as serum prolactin levels greater than 25 ng/mL)
* Cushing's syndrome
* Nonclassical congenital adrenal hyperplasia (defined as serum 17-hydroxyprogesterone levels greater than 1.2 and 5.2 ng/mL in the follicular and luteal phase, respectively) and current or previous (within the last three months) use of oral contraceptives and other hormonal
* Antidiabetic and antiobesity drugs.

Ages: 12 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Will be performed case-control study with women with Polycystic Ovary Syndrome, according to the Rotterdam criteria and body mass index between 18 to 29.9. The control group will consist of women without Polycystic Ovary Syndrome, with a body mass index of 18 to 29.9 and no other comorbidities.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Metabolic profile | 12 months
  total cholesterol (mg/dL) and fractions, triglycerides (mg/dL) will estimate

SECONDARY OUTCOMES:
Classical glycemic index | 12 months
  Classical glycemic index (mg/dL) will estimate
Liver function | 12 months
  Liver function (U/L) will estimate
luteinizing hormone | 12 months
  luteinizing hormone (IU/L) will estimate
Hormonal profile - insulin | 12 months
  Hormonal profile - insulin (uIU/ml) will estimate
Follicle stimulating hormone | 12 months
  Follicle stimulating hormone (IU/L) will estimate
thyreostimulating hormone | 12 months
  thyreostimulating hormone (uIU/ML) will estimate
Total and free testosterone | 12 months
  Total and free testosterone (ng/ml) will estimate
17-hydroxyprogesterone | 12 months
  17-hydroxyprogesterone (ng/ml) will estimate
Dehydroepiandrosterone | 12 months
  Dehydroepiandrosterone (ng/ml) will estimate
Prolactin | 12 months
  Prolactin (ug/ml) will estimate
DEXA | 12 months
  Body composition will measure by DEXA scan

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Macruz, Principal Investigator — Irmandade Santa Casa de Misericordia Sao Paulo
Locations (1):
- Carolina Furtado Macruz, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
When I have finished my recruitment and analysis of the results.

REFERENCES:
- [Derived] Macruz CF, Lima SMRR. Polycystic ovary syndrome and abdominal fat: is there a relationship? Rev Assoc Med Bras (1992). 2023 Oct 27;69(11):e20230874. doi: 10.1590/1806-9282.20230874. eCollection 2023. PMID 37909624
- [Derived] Macruz CF, Lima SM, Salles JE, da Silva GM, Scalissi NM. Assessment of the body composition of patients with polycystic ovary syndrome using dual-energy X-ray absorptiometry. Int J Gynaecol Obstet. 2017 Mar;136(3):285-289. doi: 10.1002/ijgo.12066. Epub 2017 Jan 6. PMID 28099715